CLINICAL TRIAL: NCT02074969
Title: Intramedullary Devices for the Treatment of Unstable Pertrochanteric Fractures - Epidemiological Data and Rates of Complications
Brief Title: Intramedullary Devices for the Treatment of Unstable Pertrochanteric Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Harry Widhalm, M.D., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007406
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Fractures
Keywords: re-operation rate; pertrochanteric fractures; GammaNail; PFNA; Tip-Apex-Distance; Parkers-Ratio
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gamma Nail 3 (Active Comparator): Gamma Nail 3 Stryker.
  Interventions: Device: Gamma Nail 3
- PFNA (Active Comparator): PFNA Antirotation Synthes
  Interventions: Device: PFNA

INTERVENTIONS:
Device: Gamma Nail 3 — Patients who have sustained an unstable pertrochanteric hip fracture are getting treated by Gamma Nail 3.
  Other Names: Gamma Nail 3 Stryker
  Arms: Gamma Nail 3
Device: PFNA — Patients who have sustained an unstable pertrochanteric hip fracture are getting treated by PFNA.
  Other Names: PFNA Antirotation Synthes
  Arms: PFNA

SUMMARY:
The purpose of this study is to assess the differences between two different types of devices for the treatment of unstable pertrochanteric hip fractures. The hypothesis of this study is, that patients who are treated with the proximal femoral Nail Antirotation (PFNA) have a better outcome and lower complication rates than patients treated with the Gamma Nail (GN3).

DETAILED DESCRIPTION:
This trial is a prospective randomized controlled study including the treatment of AO/OTA 31-A2 fractures in 200 patients with 2 different surgical devices. 100 patients are treated with a Gamma Nail 3 (GN3) (Stryker) the other 100 patients with a Proximal Femoral Nail Antirotation (PFNA) (Synthes).

All surgeries are performed by trauma surgeons at a Level 1 University Hospital. One hundred patients are randomized to the gamma nail and 100 are randomized to the proximal femoral nail for treatment fixation. A 1:1 randomization is performed using sealed envelopes (200 in total), which are opened by the surgeon immediately before the operation.

Patients missing an informed consent form, incomplete chart, or showing a pathologic fracture are getting excluded from final comparisons.

Patients anthropometric data as well as pre-injury mobility assessments, and ASA will be documented. Furthermore the time from admission to going to surgery, surgery length, length of stay and mobility assessment at dischargement are recorded.

After surgery the stay in the hospital is documented precisely and patients are scheduled for next appointments 2 weeks, 6 weeks, 3 months, 6 months and 1 year after surgery.

Postoperative X-rays are measured precisely to determine the Tip-Apex Distance (TAD), the Parkers-Ratio, the Singh-Score and the Neck-Shaft-Angle of the injured and contralateral side. Rates of complications as cut-out and reoperation-rates are evaluated. All intra-operative complications are noted and included in the chart.

ELIGIBILITY:
Inclusion Criteria:

* AO/OTA 31-A2 fractures
* age between 18 - 100 years
* Signed written informed consent and agreement to attend the planned FUs
* Able to understand and read country national language at an elementary level

Exclusion Criteria:

* missing informed consent form
* pathological fracture
* incomplete patient record
* death within one month of intervention (surgery)
* prior surgery to the hip
* polytrauma
* any additional fracture
* any implant at the same hip
* infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
re-operation rate | time between intervention and one year after

SECONDARY OUTCOMES:
Screw-Cut Out | time between intervention and one year after
  evaluation of sliding movements of the hip screw in the sense of a cut-out

OTHER OUTCOMES:
Mobility assessment | time between hospitalization and one year after intervention
  Mobility assessment includes scoring of pre-operative level of mobility and mobility after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Harald K. Widhalm, M.D., Principal Investigator — Department of Trauma, Medical University of Vienna, Austria
Locations (1):
- Department of Trauma, Medical University of Vienna, Vienna, Austria, Austria

REFERENCES:
- [Result] Barton TM, Gleeson R, Topliss C, Greenwood R, Harries WJ, Chesser TJ. A comparison of the long gamma nail with the sliding hip screw for the treatment of AO/OTA 31-A2 fractures of the proximal part of the femur: a prospective randomized trial. J Bone Joint Surg Am. 2010 Apr;92(4):792-8. doi: 10.2106/JBJS.I.00508. PMID 20360500